CLINICAL TRIAL: NCT03752151
Title: Micra Atrial TRacking Using A Ventricular AccELerometer 2
Acronym: MARVEL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MDT18024
Record Dates: First submitted 2018-11-14; First posted 2018-11-23 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Atrioventricular Conduction Block
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Intervention Model Description: Subjects enrolled in the MARVEL 2 study. Enrolled subjects will have the MARVEL 2 algorithm downloaded into their implanted market released Micra device. Each subject will be tested during when the MARVEL 2 algorithm is in monitor mode (VVI pacing) and in adaptive mode (VDD pacing).
Masking Description: Echocardiogram core lab will be masked to the individual patient subjects and MARVEL 2 algorithm mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MARVEL 2 Algorithm Monitor Mode, Then MARVEL 2 Adaptive Mode (Experimental): Participants first received MARVEL 2 algorithm monitor mode which provides standard VVI pacing for approximately 20 minutes followed by MARVEL 2 algorithm adaptive mode for approximately 2 hours which provides VDD pacing.
  Interventions: Device: MARVEL 2 Algorithm Monitor Mode then Adaptive Mode

INTERVENTIONS:
Device: MARVEL 2 Algorithm Monitor Mode then Adaptive Mode — Software download into implanted Micra device and programmed to MARVEL 2 Monitor Mode then MARVEL 2 Adaptive Mode

SUMMARY:
The purpose of the Micra Atrial TRacking Using A Ventricular AccELerometer 2 (MARVEL 2) study is to demonstrate safe and effective operation of the MARVEL 2 features for providing AV synchronous pacing in patients with normal sinus node function and AV block

DETAILED DESCRIPTION:
The MARVEL 2 study is an acute, prospective, global, multi-center, software-download clinical study. The study is planned to be conducted in US, Europe, and Asia. The study is expected to be conducted at approximately 15-20 centers in up to 100 subjects to obtain at least 70 usable Holter datasets to meet the objectives of the study. The expected total study duration (from first subject enrollment to the exit of the last subject) is approximately 6-months; this represents the time necessary to enroll the target sample size of at least 70 subjects with usable Holter datasets. Software will be downloaded into patients implanted with a Micra device to allow the new algorithm performance to be measured in patients where a Micra device has already been chosen as most appropriate for the patient.

Most enrolled subjects will complete the study procedures during a single study visit. However, subjects enrolling in the study at the time of their Micra implant (anticipated to be approximately 10 subjects) will have the investigational algorithm downloaded following Micra implant, prior to hospital discharge, and approximately 1-month post-implant. This subset of subjects with de novo Micra implants will allow the MARVEL 2 features to be tested at multiple points in the device life cycle.

Since the download algorithm running in a Micra device significantly increases current drain, a 2-4 hour acute study is used to limit the reduction in device longevity.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been implanted with a Micra TPS (Model MC1VR01) with remaining device longevity of 6 years or more or is expected to be implanted with a Micra TPS.
* Subject has history of AV block*
* Subject is ≥ 18 years old and as per required local law.
* Subject (and/or witness as applicable per local regulations) provides signed and dated authorization and/or consent per institution and local requirements.
* Subject is willing and able to comply with the protocol. *This includes subjects with normal sinus function and persistent 3rd degree AV block and subjects with other forms of AV block.

Exclusion Criteria:

* Subject is currently enrolled or planning to participate in a potentially confounding drug or device trial during the study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic Clinical Research Specialist.
* Subject is pregnant (if required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to MARVEL 2 study procedures).
* Subject meets any exclusion criteria required by local law (age or other).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Baptist Hospital, Miami, Florida
  - North Shore University Hospital- Northwell, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
- Kepler Universitätsklinikum Med Campus III, Linz, Austria
- UZ Leuven - Campus Gasthuisberg, Leuven, Belgium
- Odense Universitetshospital, Odense C, Denmark
- Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac, France
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Hospital Universitari Clínic de Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Garweg C, Khelae SK, Chan JYS, Chinitz L, Ritter P, Johansen JB, Sagi V, Epstein LM, Piccini JP, Pascual M, Mont L, Willems R, Splett V, Stromberg K, Sheldon T, Kristiansen N, Steinwender C. Behavior of AV synchrony pacing mode in a leadless pacemaker during variable AV conduction and arrhythmias. J Cardiovasc Electrophysiol. 2021 Jul;32(7):1947-1957. doi: 10.1111/jce.15061. Epub 2021 May 20. PMID 33928713
- [Derived] Garweg C, Khelae SK, Steinwender C, Chan JYS, Ritter P, Johansen JB, Sagi V, Epstein LM, Piccini JP, Pascual M, Mont L, Willems R, Sheldon T, Splett V, Stromberg K, Wood N, Chinitz L. Predictors of atrial mechanical sensing and atrioventricular synchrony with a leadless ventricular pacemaker: Results from the MARVEL 2 Study. Heart Rhythm. 2020 Dec;17(12):2037-2045. doi: 10.1016/j.hrthm.2020.07.024. Epub 2020 Jul 24. PMID 32717315
- [Derived] Steinwender C, Khelae SK, Garweg C, Chan JYS, Ritter P, Johansen JB, Sagi V, Epstein LM, Piccini JP, Pascual M, Mont L, Sheldon T, Splett V, Stromberg K, Wood N, Chinitz L. Atrioventricular Synchronous Pacing Using a Leadless Ventricular Pacemaker: Results From the MARVEL 2 Study. JACC Clin Electrophysiol. 2020 Jan;6(1):94-106. doi: 10.1016/j.jacep.2019.10.017. Epub 2019 Nov 11. PMID 31709982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were considered enrolled when they signed informed consent Subjects were enrolled between 22 January 2019 and 14 June 2019 at 12 study centers in 8 countries
Pre-assignment Details: Following enrollment, the MARVEL 2 algorithm was downloaded into the subject's implanted Micra pacemaker. Following download subjects were programmed to MARVEL 2 Algorithm monitor mode followed by MARVEL 2 adaptive mode. Two subjects exited prior to MARVEL 2 download; one did not meet the study inclusion/exclusion and one withdrew consent.
Groups:
- MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode: Participants were programmed to MARVEL 2 algorithm monitor mode which provides standard VVI pacing for approximately 20 minutes. Then the MARVEL 2 algorithm was programmed to adaptive mode which provides VDD pacing for approximately 2 hours.
Period: Overall Study
Arm/Group | MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode
Started | 77
Completed | 75
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The baseline population is the number of participants who signed the study's informed consent
Groups:
- MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive: Participants were programmed to MARVEL 2 algorithm monitor mode which provides standard VVI pacing for approximately 20 minutes. Then the MARVEL 2 algorithm was programmed to adaptive mode which provides VDD pacing for approximately 2 hours.
Arm/Group | MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One patient who withdrew prior to download of the MARVEL 2 algorithm did not complete the baseline procedures.
  years
    number analyzed (Participants) | 76
    (all) | 77.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient who withdrew prior to download of the MARVEL 2 algorithm did not complete the baseline procedures.
  Participants
    number analyzed (Participants) | 76
    Female | 31
    Male | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 6
  Belgium | 20
  Hong Kong | 11
  United States | 14
  Denmark | 4
  Malaysia | 15
  France | 6
  Spain | 1
Predominant heart rhythm [Count of Participants; unit: Participants] — Predominant heart rhythm as assessed on electrocardiogram during Holter monitoring
  Participants
    Persistent 3rd degree AV block with normal sinus | 40
    Intact atrioventricular conduction | 18
    Other rhythm | 15
    Rhythm indeterminate | 2
    Participant exited prior to software download | 2

OUTCOME MEASURES:

1. Primary Outcome: Atrial Ventricular Pacing Synchrony Success During Rest
Description: A subject will meet the primary endpoint if a paced or sensed ventricular beat is within 300 ms following an ECG confirmed P-wave for at least 70% of the ECG confirmed P-waves. The primary endpoint will be evaluated during the MARVEL 2 setup phase during MARVEL 2 Algorithm monitor mode (VDI pacing which is effectively VVI pacing) and during the 20-minute resting period in which the MARVEL 2 Algorithm is programmed to Adaptive mode (VDD pacing)
Time Frame: 40 Minutes
Population: Participants with a predominant heart rhythm of 3rd degree atrioventricular block and normal sinus function during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive
Number analyzed (Participants) | 40
Participants
  Monitor Mode Success and Adaptive Mode Success | 0
  Monitor Mode Failed and Adaptive Mode Success | 38
  Monitor Mode Success and Adaptive Mode Fail | 0
  Monitor Mode Fail and Adaptive Mode Fail | 2
Statistical Analysis 1: Comparison: MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive; The null hypothesis was that the probability of meeting the endpoint (Atrioventricular synchrony >70%) was the same in MARVEL 2 Monitor Mode and MARVEL 2 Adaptive Mode. A sample size of 35 participants with a predominant rhythm of 3rd degree atrioventricular block and normal sinus function provided >90% power at a type I error rate of 0.05 assuming the proportion of patients meeting the endpoint in one mode, but not the other exceeded 50% and 90% of these pairs favored the Adaptive mode; Test type: Superiority; p < 0.001, McNemar

2. Primary Outcome: Number of Participants Free From Inappropriate Pacemaker Function Events
Description: A participant will meet the primary endpoint if they are free from the following MARVEL 2 software related events during the entire Holter monitoring period where the MARVEL 2 features are enabled.
  Inappropriate pacemaker function events are defined as:
  1. Cardiac pauses lasting longer than 2 cardiac cycles (where cardiac cycle length is defined by the programmed lower rate interval of the pacemaker), OR
  2. Pacemaker oversensing induced tachycardia exceeding 3-minutes, defined as oversensing of the pacemaker's accelerometer signal leading to a heart rate exceeding 100 beats per minute.
Time Frame: Through study completion an average of one day
Population: Number of participants with the MARVEL 2 software downloaded onto their Micra implanted pacemaker
Measure: Count of Participants; unit: Participants
Arm/Group | MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode
Number analyzed (Participants) | 75
Participants | 75
Statistical Analysis 1: Comparison: MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode; The null hypothesis is that 87% or fewer participants will achieve the endpoint. The alternative hypothesis is that more than 87% of participants will achieve the endpoint. A sample size of 70 participants provides at least 90% power to test the null hypothesis assuming the true rate of meeting the endpoint in the population is 98% at a type I error rate of 2.5%; Test type: Superiority; p < 0.001, Exact binomial test; proportion expressed as a percentage = 100, 95% CI 2-sided [95.2 to 100]

3. Secondary Outcome: Left Ventricular Outflow Tract Velocity Time Integral
Description: The secondary endpoint is left ventricular outflow tract (LVOT) velocity time integral (VTI) as obtained from echocardiogram while the MARVEL 2 features are in adaptive mode (VDD pacing) and while the MARVEL 2 features are in monitor mode (VDI pacing which is effectively VVI pacing). This was measured by the echo core laboratory that was blinded to the study participant and MARVEL 2 algorithm mode.
Time Frame: 12 cardiac cycles
Population: Participants with paired LVOT VTI measurements during MARVEL 2 Adaptive mode (VDD pacing mode) and MARVEL 2 Monitor mode (VDI pacing which is effectively VVI pacing) with a predominant heart rhythm of persistent 3rd degree atrioventricular block and normal sinus rhythm
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode
Number analyzed (Participants) | 39
cm | 1.7 [0.7 to 2.7]
Statistical Analysis 1: Comparison: MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode; The null hypothesis is that the mean LVOT VTI during MARVEL 2 Adaptive mode equals the mean LVOT VTI during MARVEL 2 Monitor mode. A sample size of 35 participants with paired LVOT VTI measurements provides 89% power at a type I error rate of 5% to reject the null hypothesis assuming the true difference in LVOT VTI is 2.1 cm with a standard deviation of 3.8 cm; Test type: Superiority; p = 0.002, t-test, 2 sided; Paired t-test since each participant had LVOT VTI measurements in MARVEL 2 Adaptive and Monitor modes; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [0.7 to 2.7]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 3/75
Other Adverse Events (participants affected / at risk) | 3/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode (N=75)
Hypotension (Vascular disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Myocardial haemorrhage (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MARVEL 2 Monitor Mode Then MARVEL 2 Adaptive Mode (N=75)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, the contract allows the principal investigator to publish their data after release of a multi-center publication per the publication strategy following Medtronic's review for disclosure of confidential information ("CI"), technical correctness, disclosure of patentable or copyrightable material, and selection and order of publications by the publications committee. Any such CI and/or item identified as not technically correct is deleted prior to publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT03752151/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT03752151/SAP_001.pdf